CLINICAL TRIAL: NCT07069478
Title: Cannabidiol (CBD) and Stress Response: Psychobiological Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DMED-2025-33636
Record Dates: First submitted 2025-05-28; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: CBD; Cannabidiol; Stress; Acute Stress Reaction
Keywords: cardiovascular reactivity, , , ,; hypothalamic-pituitary-adrenal axis; stress; mood; CBD use
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Single group assignment; all participants experience baseline rest, acute stress tasks, and recovery rest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants will include CBD users and non users
  Interventions: Other: Stress Intervention

INTERVENTIONS:
Other: Stress Intervention — Experimental Stress: Behavioral induction of acute psychosocial and physiological stress. First, participants will be provided with a speech topic and given 4 minutes to prepare a speech that they subsequently deliver in front of evaluators and a video recorder. Then, participants will complete a mental arithmetic task in front of the evaluators for 8 minutes. Then, participants will complete a cold pressor task in which they submerge their hand in ice water for 90 seconds.

SUMMARY:
The aim of this study is to determine the effects of regular cannabidiol (CBD) use on the psychobiological mechanisms of the stress response. This will be achieved by comparing acute stress responses of adults who either use or do not use CBD regularly. Correlates of CBD use, including tobacco use, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are relatively healthy and aged 21-70 years.
* Must keep a normal sleep schedule (sleep during nighttime, awake during daytime).
* Must either (1) use CBD daily/regularly or (2) not use CBD regularly.

Exclusion Criteria:

* Participated in previous acute stress studies that included a similar stress induction.
* Current, unstable: major psychiatric disorder or medical condition (e.g., uncontrolled hypertension above 160/100).
* Self-reported current pregnancy.
* Self-reported current use of illicit substances (other than cannabis).
* Non-compliance with instructions for study visit (abstinence from alcohol, caffeine, physical activity, etc.)
* Students of the principal researcher

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in subjective states (stress, anxiety, positive affect) | 2.5 hours
  Participants will self-report the extent to which they have felt stressed, overwhelmed, anxious/nervous, cheerful, and happy during the last 30 minutes before acute stress, immediately after acute stress, and after a recovery period. The Subjective States Questionnaire will be used to score responses. The minimum values are 0 (not at all) and the maximum values are 7 (very strongly). Higher scores mean more stress, more anxiety, and more positive affect.
Change in cardiovascular activity and cortisol | 2.5 hours
  Saliva will be collected (for later cortisol assays) and cardiovascular activity will be measured before, during, and after acute stress.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa al'Absi, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States